CLINICAL TRIAL: NCT05482061
Title: Predictors of Treatment Failure Pain Among Patients Gunshot Wounds
Acronym: PTFPAPGW
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Principal Investigator, Bogomolets National Medical University
Other Study IDs: №158, 23.05.2022
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury. The basic tool for pain intensity research was the VAS. The study of the neuropathic component of pain was carried out using the DN4. Study of the presence of an acute stress reaction - anamnesis + HADS. The diagnosis of ASR was established by a psychiatrist upon admission to the military mobile hospital. The presence of post-traumatic stress disorders (PTSD) was investigated using the Mississippi scale of post-traumatic stress disorders (military version). The presence of PTSD according to the MS PTSD (c). Satisfaction with treatment results was studied using the Chaban Quality of Life Scale.
  Interventions: Other: visual analog scale (VAS).
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv. All patients who took part in the study with gunshot wounds were evacuated to the stage of treatment - the National Military Medical Clinical Center "Main Military Clinical Hospital". The research was conducted using the same methods as during the retrospective analysis. The exception is the study period during treatment at the military medical clinical center: here it was 14 days.
  In all patients with gunshot wounds, the outcome and effectiveness of pain management were assessed using the Visual Analogue Scale (VAS) and the Diagnostic Questionnaire for the Detection of the Neuropathic Pain Component Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36 (DN4).
  Interventions: Other: visual analog scale (VAS).

INTERVENTIONS:
Other: visual analog scale (VAS). — The basic tool for pain intensity research was the VAS: 1) before and after anesthesia - at the stage of the medical and nursing brigade, military mobile hospital, military medical clinical center; 2) at the stage of the medical and nursing team - within 2 days; 3) at the stage of the military mobile hospital - within 5 days; 4) at the stage of the military medical clinical center - within 7 days, at the time of discharge from the hospital; 5) at the rehabilitation stage. Intervals between analgesia were also studied. The study of the neuropathic component of pain was carried out using the diagnostic DN4: military mobile hospital, a military medical clinical center, then at the time of discharge from a military medical clinical center. Study of the presence of an acute stress reaction - anamnesis + The Hospital Anxiety and Depression Scale. Satisfaction with treatment results was studied using the Chaban Quality of Life Scale.
  Other Names: neuropathic pain Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36 (DN4).; The Hospital Anxiety and Depression Scale (HADS); Mississippi scale of post-traumatic stress disorders (military version); Satisfaction with treatment results was studied using the Chaban Quality of Life Scale

SUMMARY:
In patients with gunshot wounds during hostilities in Ukraine, 76.9% have negative results of pain treatment, which leads to its chronicity. Identifying predictors of negative pain outcomes in these patients may improve their treatment outcomes.

DETAILED DESCRIPTION:
One of the strongest factors that has a psychological impact on a person is war and conditions in which injury occurs, conditions in which pain occurs. A gunshot wound received during the war in the conditions of hostilities becomes the reason for the indisputable association of pain sensations with the events in which the patient was injured. It is pain and memories, memories and pain that cause the development of states with self-destructive behavior. According to statistics, gunshot wounds account for 54-70%. Gunshot wounds to the chest during anti-terrorist operations/OOS make up 7.4-11.7%, shrapnel wounds prevail here - 72.2%, explosive wounds - 17.5%, bullet wounds - 10.3%, and lethality - 12.2 -25%. According to the data of the Command of the Medical Forces of the Armed Forces of Ukraine, in the structure of gunshot injuries, 64% are injuries to the limbs: of them, 74.8% are soft tissues, 25.2% are gunshot fractures, bone defects are noted in 11.6% of patients, and wounded.

The study of predictors of negative results of pain treatment in patients with gunshot wounds requires in-depth study, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions have their own characteristics. Since in 76.9% of cases it is not possible to achieve a positive result of treatment, the data of our study will play an important role in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* presence of gunshot wounds during hostilities, male gender

Exclusion Criteria:

* absence of gunshot wounds during hostilities, other sex

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1049 patients with gunshot wounds during hostilities were retrospectively studied. 1166 patients with gunshot wounds during hostilities were prospectively studied
Sampling Method: Non-Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  from 0 to 10 points (the intensity of pain is determined)
Didier Bouhassiraa DN4 | 12 months
  the number of points 4 or more indicates that the patient has a neuropathic pain component
The Hospital Anxiety and Depression Scale | 12 months
  more than 7 points indicates the presence of anxiety/depression
Mississippi PTSD scale (military version) | 12 months
  average values of the total score are 76±18 for well-adjusted servicemen, 86±26 for servicemen with mental disorders, 130±18 for PTSD
Chaban Quality of Life Scale | 12 months
  assesses quality of life and satisfaction with treatment results up to 56 points - very low 57-66 - low 67-75 - average 76-82 - tall 83-100 is very high

CONTACTS AND LOCATIONS:
Overall Officials: Vasyl' Horoshko, PhD, Principal Investigator — Bogomolets National Medical University, Ministry of Health of Ukraine
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No